CLINICAL TRIAL: NCT06112106
Title: A Multi-center, Randomized, Parallel-group, 4-month Study to Compare the Effect of Ergonomic Recommendations Versus Intelligent Physical Exercise Training (IPET) and Ergonomic Recommendations on Musculoskeletal Pain Among Abdominal and Pelvic Surgeons.
Brief Title: The Effect of Intelligent Exercise and Ergonomic Recommendations on Surgeon Musculoskeletal Discomfort
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Working Environment Research Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20205100734
Record Dates: First submitted 2023-10-04; First posted 2023-11-01 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2024-08

CONDITIONS: Occupational Injuries; Occupational Exposure
Keywords: Ergonomics; Physical exercise training; Prevention; Rehabilitation; Microbreaks; Surgeons
MeSH Terms: conditions — Occupational Injuries

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigator who performs the statistical analysis will be masked to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Surgeons assigned to the control group will be asked (to continue) to apply the ergonomic recommendations in the daily practice introduced three months ahead of trial start.
- Intervention group (Experimental): Surgeons
  Interventions: Behavioral: Intelligent Physical Exercise Training (IPET)

INTERVENTIONS:
Behavioral: Intelligent Physical Exercise Training (IPET) — The intervention group will follow an Intelligent Physical Exercise training (IPET) program delivered via a mobile phone app. The scope of the physical exercise program is 50 minutes per week, and it is individually tailored according to questionnaire responses about work profile, physical capacity, health status and extent of musculoskeletal pain.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to investigate the effects of Intelligent Physical Exercise Training (IPET) and ergonomic recommendations on musculoskeletal pain among abdominal and pelvic surgeons. The main question it aims to answer is:

• Is IPET superior to ergonomic recommendations in rehabilitating or preventing musculoskeletal pain?

12 weeks ahead of trial start, all participants will be familiarized with ergonomic principles in the operating room. In the 20-week trial, the control group is asked to resume practicing and applying the ergonomic principles when they operate. In addition to applying the ergonomic principles, the Intervention group will be asked to perform 50 min. per week of individually tailored physical exercise training. The program is delivered via an application (app).

DETAILED DESCRIPTION:
Pre-intervention The three months leading up to the trial start, all participants are introduced to up-to-date ergonomic recommendations. The ergonomic recommendations are informed by general ergonomic recommendations from the Danish Working Environment Authority, a systematic literature review on the effect of ergonomic interventions applied in the OR (REF and general ergonomic guidelines) and include two recommendations: 1) performing intra-operative microbreaks, and 2) knowledge of ergonomic work posture in the OR.

InterventionIntelligent Exercise app + ergonomic recommendations The duration of the ergonomic recommendations launch period is three months after which consenting participants will be randomized to either the control group or the intervention group. The control group will be encouraged to continue to apply the up-to-date ergonomic recommendations to their OR practice, this will act as usual care. In addition to the usual care, the intervention group will be prescribed individualized physical exercise training (IPET). The IPET is 50 min of tailored physical exercise per week, that is designed by an algorithm that uses the information (demographics, self-reported health, musculoskeletal pain and its location) the individual enters in the app (REF). The 50 min. Of total IPET per week can be performed in one session or divided into shorter sessions two-five sessions with the same effect (REF). The IPET will be delivered through the participants' mobile phone via a mobile application (app) that requires a unique code assigned for each participant. Each participant's exercise training program is different because it is composed of the input provided by the participant. Thus, as the participants experience progress (or deterioration) in their physical capacity during the study, the program will change accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Surgeon in gynecologic-, urologic, colorectal or abdominal surgery
* Performs an average of four hours of surgery per week

Exclusion Criteria:

* Own physician has advised against performing physical exercise training

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Musculoskeletal pain intensity | Assessed at baseline (pre-intervention), 12 weeks and 20 weeks (post-intervention)
  Pain intensity on a 11-point Likert scale (0= no pain, 10= most intense pain) the past 3 months and last 7 days in neck, shoulders, elbows/arms, wrists/hands, upper back, lower back, hips, knees, ankle/feet

SECONDARY OUTCOMES:
Self-reported use of pain medicine | Assessed at baseline (pre-intervention), 12 weeks and 20 weeks (post-intervention)
  Use of pain medicine due to musculoskeletal pain. Answer categories: daily, one to several times a week, one to several times a month, rarely or never
Self-reported time spent on moderate to vigorous physical activity during a regular week (in minutes) | Assessed at baseline (pre-intervention), 12 weeks and 20 weeks (post-intervention)
  Accumulated physical activity during a regular week (hours/minutes). Answer categories for moderate physical activity: less than 30 min., 30-90 min., 90-149 min., 150-299 min., 300 min. or more. Answer categories for vigorous physical activity: less than 30 min, 30-89 min, 90-149 min, 150 min. or more.
Self-reported physical resources | Assessed at baseline (pre-intervention), 12 weeks and 20 weeks (post-intervention)
  Rating own physical resources (cardiorespiratory fitness, strength, balance) compared to peers on a Likert scale (0= poor, 10= good).
Self-reported health | Assessed at baseline (pre-intervention), 12 weeks and 20 weeks (post-intervention)
  General health answer categories: On a five-point Likert scale (0= excellent, 5= poor). Physical and mental health rated on various likert scales.
Self-reported personal and work-related burnout | Assessed at baseline (pre-intervention), 12 weeks and 20 weeks (post-intervention)
  The Copenhagen Burnout Inventory. Answer categories: 5-point Likert scales from "always" to "almost never or never", or from "very much" to "very little"
Self-reported work ability | Assessed at baseline (pre-intervention), 12 weeks and 20 weeks (post-intervention)
  The Work Ability Index (WAI) contains questions concerning work, work ability and health.
Working conditions | Assessed at baseline (pre-intervention), 12 weeks and 20 weeks (post-intervention)
  Surgical specialty, weekly workings hours as primary and assisting surgeon
Musculoskeletal pain frequency past 3 months | Assessed at baseline (pre-intervention), 12 weeks and 20 weeks (post-intervention)
  Pain frequency for the past 3 months (possible answers: 0d, 1 to 7d, 8 to 30d, more than 30 days but not every day, every day)

CONTACTS AND LOCATIONS:
Overall Officials: Helle J Christiansen, Msc., Principal Investigator — University of Aarhus
Locations (7):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
- Denmark (5):
  - Aarhus University, Aarhus
  - Gødstrup Regional Hospital, Gødstrup
  - Odense University Hospital, Odense
  - Randers Regional Hospital, Randers
  - Sygehus Lillebælt, Vejle, Vejle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christiansen HJ, Sandal LF, Mogensen O, Norasi H, Chrouser K, Hallbeck MS, Jensen PT, Dalager T. Prevention and rehabilitation of musculoskeletal pain among abdominal and pelvic surgeons with intelligent physical exercise training (IPET) and intraoperative ergonomic recommendations (ERGO): study protocol for a multicenter open-label randomized controlled trial in Denmark and North America (USA). Trials. 2025 Dec 12;26(1):565. doi: 10.1186/s13063-025-09178-x. PMID 41388556